CLINICAL TRIAL: NCT06696339
Title: Collection of Fingertip Video for Determination of Heart Rate
Brief Title: Assessment of Heart Rate Measurement Accuracy for the PreemptiveAI SDK in Adults
Status: Active, not recruiting | Type: Observational
Sponsor: PreemptiveAI, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: HR-001
Record Dates: First submitted 2024-10-23; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Heart Rate in the General Public

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: PreemptiveAI SDK — Use the PreemptiveIAI SDK to measure heart rate.

SUMMARY:
The goal of this clinical trial is to assess the accuracy of the PreemptiveAI SDK to measure heart rate for adults as compared to an FDA-approved ground truth device.

Participants will:

* Complete a demographics and health history survey
* Apply and wear ground truth equipment such as a pulse oximeter and ECG
* Measure their heart rate 8 times with 4 different smartphones using the PreemptiveAI SDK

ELIGIBILITY:
Inclusion Criteria:

* Adults with both normal and abnormal heart rates

Exclusion Criteria:

* Under 18 years of age
* Unable to speak and read English
* Deemed not suitable to participate by Investigator due to cognitive impairment, acute illness, or serious physical or mental health condition
* Essential tremor in left or right hand
* Raynaud's disease
* Severe calluses on left or right index finger
* Unable to produce a heart rate measurement due to low signal quality during the training phase (i.e. low perfusion, unable to hold hand steady, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: At least 60 participants, up to 125 participants. Participants will be recruited to meet the following demographics goals:
  * Sex assigned at birth - a minimum of 25 male and 25 female participants
  * Age - a minimum of 10 participants in each age bin: 18-30, 30-65, 65+
  * BMI - a minimum of 5 participants in each bin: 0-25, 25-30.0, 30.0+
  * Skin tone (Fitzpatrick scale) - a minimum of 10 participants in each bin: Type 1/2, Type 3/4, Type 5/6
  * Heart Rate - a minimum of 5 participants with average heart rate < 60 bpm and >100 bpm
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Error | At single site visit, measured across 8 repetitions within a 1-hour period
  Root mean square error of heart rate compared to ground truth device

CONTACTS AND LOCATIONS:
Locations (1):
- Paul Allen Institute for Artificial Intelligence, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No